CLINICAL TRIAL: NCT04126850
Title: Pilot Project: The Amplicon and Metatranscriptomic Next-generation Sequencing of Samples From Intra and Extra-intestinal Microbiome in Non-infectious Uveitis Patients to Decipher Possibility Uveitis Pathogenesis
Brief Title: Pilot Project: The Amplicon and Metatranscriptomic Study of Intra and Extra Intestinal Microbiome in Non-infectious Uveitis Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, Ratna Sitompul, Prof. Dr. dr. Ratna Sitompul, SpM(K), Fakultas Kedokteran Universitas Indonesia
Other Study IDs: 19-05-0624
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Autoimmune Uveitis; Behçet Disease; Vogt-Koyanagi-Harada Disease; Idiopathic Uveitis; Noninfectious Panuveitis; Anterior Uveitis Idiopathic; Posterior Uveitis; Intermediate Uveitis
Keywords: Microbiome; Autoimmune Uveitis; Vogt-Koyanagi-Harada Disease; Behçet Disease; Idiopathic Uveitis; Metatranscriptomic; Amplicon
MeSH Terms: conditions — Behcet Syndrome; Uveomeningoencephalitic Syndrome; Uveitis, Posterior; Uveitis, Intermediate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Feces
  * Blood
  * Aqueous humor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to discover the composition on the microbiome in several sites of the human body; and to find out the difference in microbiome composition on ocular fluid, blood, and feces before and after therapy in uveitis patient with history of autoimmune disease (Behcet and Vogt-Koyanagi-Harada) and idiopathic uveitis

DETAILED DESCRIPTION:
Gut microbiome has been widely studied around the globe, and it is convinced that the gut microbiome plays an essential role in many human diseases. In a published review showed the presence of microbes in blood from a patient who suffered from non-communicable disease. The microbes present in dormant or not-immediately-culturable states as if blood is a 'sterile' environment. It was argued that the difficulty of culturing microbes from the blood was coming from the limited understanding of suitable growth/isolation media for the microbes to be cultured. This limitation can be overcome by the sequenced-based methods for detecting non-proliferating microbes. The presence of microbes in blood also can be observed by ultrastructural (microscopic) methods. Through the microscopic observations, it was witnessing the presence of coccus and bacillus shaped bacteria that present proximity to (Red Blood Cell) RBCs in sample blood patients with Alzheimer's or Parkinson's Disease. The presence of microbes in the places other than their normal location state by term 'atopobiosis'. The presence of microbes in blood suspected as a result of translocation between the gut to the blood.

Therefore, according to the current knowledge of microbiome association and the human diseases, we are eager to conduct a pilot project that gives a comprehensive picture of the association between the microbiome and uveitis disease partially non-infectious and idiopathic uveitis. We will investigate microbiome profiling in the intestinal and extra-intestinal of uveitis patients before and after treatment to see whether any alteration of microbial abundance at two distinct clinical conditions partially in uveitis patients with history of autoimmune disease (Behcet and Vogt-Koyanagi-Harada) and idiopathic uveitis. Another objective of this study is to explore any pathogenic microorganism that present in uveitis patients samples conducted by a sequenced-based method.

ELIGIBILITY:
Inclusion Criteria:

* New patient registered at Cipto Mangunkusumo Hospital since November 2019
* Patient diagnosed with non-infectious uveitis (with Behcet, VKH history)
* Patient idiopathic uveitis (proven to have negative result by available etiological uveitis work-ups)
* Minimum age: 18 years old
* Experience active inflammation in the past 180 days and or during patient registration following Standard Uveitis Nomenclature (SUN) guidelines, in at least:

  * equal and or more than 2+ anterior chamber cells
  * equal and or more than 2+ vitreous haze and/or
  * active retinal/choroidal lesions

Exclusion Criteria:

* patients had taken probiotics supplement or antibiotics 3 months before sample collection
* or who experience prolonged diarrhea or constipation
* or undergone gastrointestinal surgery
* having any form of malignancy
* having a systemic disease such as hypertension, obesity, inflammatory bowel disease, or diabetes.
* Disagree to sign informed consent
* Uveitis is proven to be an infectious origin
* Pregnant patient
* Loss to follow up patient

Healthy volunteers are recruited for this study after giving consent with the following inclusion criteria:

* age: 18-50 years old (Man/Woman)
* having no health complaints or symptoms
* not in any long term medications
* having no history of allergy
* willing to cooperate in the study
* state of complete physical, mental and social well being

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Non-infectious and idiopathic uveitis patients registered from November 2019 at Cipto Mangunkusumo Hospital, Indonesia.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Differential abundant taxonomic groups bacterial | 0, 6 weeks
  The primer used in this amplicon study is targeted to 16S rRNA gene region V3-V4 to detect bacterial diversity in the samples. The sequencing will be generated by Illumina according to standard protocol. Prior filter is conducted using Prinseq-lite, then chimeric sequences remove using Usearch61 and left over the high quality reads. The (operational taxonomic unit) OTU is picked using bioinformatic tool (Quantitative Insights Into Microbial Ecology - QIIME). Taxonomic classification for de novo OTUs clustering will be generated using open source software package for bioinformatics data processing. Shanon diversity, Simpson index will be examined for calculating alpha diversity. And then we will do identification of differential abundant taxonomic groups. And do analysis correlation network between bacterial genera among two clinical condition (before and after received oral steroid) relatively to health control.

SECONDARY OUTCOMES:
Detection pathogenic microorganism in samples | 0, 6 weeks
  In this study we are going to use IDseq Portal, a novel bioinformatics platform that designed for detection of microbes from metagenomic data. This analysis will be applied in all types samples (stool, blood, and aqueous humor). We expect to find any specific microbiome (bacterial/fungal/virus) signature in samples patient uveitis.

CONTACTS AND LOCATIONS:
Overall Officials: Ratna Sitompul, Professor, Principal Investigator — RSUPN dr. Cipto Mangunkusumo Hospital (RSCM)
Locations (1):
- RSUPN dr. Cipto Mangunkusumo (Cipto Mangunkusumo Hospital), Jakarta Pusat, Jakarta Special Capital Region, Indonesia